CLINICAL TRIAL: NCT06462456
Title: Post-market Clinical Follow-up Study of Alcon PRECISION1™ Spherical Soft Contact Lenses (Verofilcon A) and PRECISION1T™ for Astigmatism Contact Lenses (Verofilcon A)
Brief Title: Post-market Clinical Follow-up Study of Alcon PRECISION1™ Spherical and PRECISION1™ for Astigmatism Soft Contact Lenses
Status: Terminated | Type: Observational
Why Stopped: Management decision
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Other Study IDs: CLE383-I001
Record Dates: First submitted 2024-06-12; First posted 2024-06-17 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Refractive Errors
Keywords: Myopia; Hyperopia; Astigmatism
MeSH Terms: conditions — Refractive Errors; Myopia; Hyperopia; Astigmatism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- PRECISION1 Sphere: Verofilcon A spherical soft contact lenses worn in both eyes in a real-world setting
  Interventions: Device: Verofilcon A spherical soft contact lenses
- PRECISION1 Toric: Verofilcon A toric soft contact lenses worn in both eyes in a real-world setting
  Interventions: Device: Verofilcon A toric soft contact lenses

INTERVENTIONS:
Device: Verofilcon A spherical soft contact lenses — Silicone hydrogel contact lenses prescribed for single use, daily disposable wear (less than 24 hours while awake) for the correction of ametropia (myopia or hyperopia)
  Other Names: PRECISION1™
  Groups: PRECISION1 Sphere
Device: Verofilcon A toric soft contact lenses — Silicone hydrogel contact lenses prescribed for single use, daily disposable wear (less than 24 hours while awake) for the correction of ametropia (myopia or hyperopia) with astigmatism
  Other Names: PRECISION1™ for Astigmatism
  Groups: PRECISION1 Toric

SUMMARY:
The purpose of this study is to assess long term performance and safety of verofilcon A soft contact lenses in a real-world setting in a population of 7 years or older having at least 1 year of verofilcon A (sphere or toric) contact lens wear in a daily wear and daily disposable modality.

DETAILED DESCRIPTION:
This study consists of a Baseline Visit and a Year 1 Visit.

The Baseline Visit is defined as the first office visit where an eye care professional provided an in-person office biomicroscopy exam to the subject before or during which a PRECISION1™ sphere or toric contact lens prescription was released. The Baseline Visit will be retrospective, with all assessments obtained from chart review.

The Year 1 Visit is defined as the visit that occurs 1 year (-2/+4 months) since Baseline during which period the subject is wearing test lenses of the same design in both eyes and a contact lens examination is performed during the visit. The Year 1 Visit may be prospective or retrospective.

ELIGIBILITY:
Key Inclusion Criteria:

* Subject (or subject's legal representative) is able to understand and sign an informed consent/assent form approved by an Institutional Review Board (IRB), unless appropriate consent waiver for the retrospective chart review is provided by the IRB.
* Verofilcon A (sphere or toric) contact lens wear as described in the protocol.
* Best corrected spectacle distance visual acuity (VA) 20/25 or better at baseline.
* Healthy, non-diseased eyes, as determined/known by the Investigator.
* Other protocol-defined inclusion criteria may apply.

Key Exclusion Criteria:

* Any ocular disease or condition that would contraindicate contact lens wear present at baseline.
* Use of systemic or ocular medications that would contraindicate contact lens wear at baseline.
* Other protocol-defined exclusion criteria may apply.

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects will be recruited from clinical sites located in the United States.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2024-08-30 (Actual); Primary Completion 2025-03-11 (Actual); Study Completion 2025-03-11 (Actual)

PRIMARY OUTCOMES:
Distance Visual Acuity with Study Lenses at Baseline | Baseline
  Visual acuity (VA) assessed per the investigator's standard of care with study lenses in place.
Distance Visual Acuity with Study Lenses at Year 1 Follow-Up | Year 1
  Visual acuity (VA) assessed per the investigator's standard of care with study lenses in place.
Incidence of Corneal Infiltrative Events | Up to Year 1
  A corneal infiltrate is a single or group of inflammatory cells in the normally clear cornea.
Incidence of Microbial Keratitis | Up to Year 1
  Microbial keratitis is a sight-threatening infection of the cornea.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Lead, VC, Study Director — Alcon Research, LLC
Locations (12):
- United States (12):
  - Scripps Optometric Group, San Diego, California
  - Pearle Vision, Jacksonville, Florida
  - Vision Health Institute, Orlando, Florida
  - Vision Salon Eye Care Associates, Blue Island, Illinois
  - Illinois College of Optometry, Chicago, Illinois
  - CORL, Indiana University, Bloomington, Indiana
  - The Eye Doctors Inc, Eden Prairie, Minnesota
  - Cornea and Contact Lens Institute of Minnesota, Edina, Minnesota
  - Complete Eye Care of Medina, Medina, Minnesota
  - Spectrum Eyecare, Jamestown, New York
  - Eyecare Professionals, Inc, Powell, Ohio
  - Optometry Group, PLLC, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: No